CLINICAL TRIAL: NCT03810235
Title: Transdermal Lidocaine Patch for Post-Cesarean Pain Control for Women With Obesity: a Single-blind Randomized Controlled Trial
Brief Title: The OBstetric Lidocaine Patch (OBLido) Trial
Acronym: OBLido
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Meriter IRB 2018-015; A532860 (Other: UW Madison); SMPH/OBSTET & GYNECOL/OBSTET (Other: UW Madison); 2019-0139 (Other: UW-Madison IRB)
Record Dates: First submitted 2019-01-07; First posted 2019-01-18 (Actual); Results first posted 2020-09-07 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2022-10

CONDITIONS: Pain, Postoperative
Keywords: lidocaine; patch
MeSH Terms: conditions — Pain, Postoperative | interventions — Bandages, Hydrocolloid

STUDY DESIGN:
Intervention Model Description: single-center, single blind, randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Transdermal Lidocaine Patch (Active Comparator): Drug: Including placebo The intervention is the post-operative application of a 5% lidocaine transdermal patch for women who have undergone Cesarean delivery.
  Interventions: Drug: Transdermal Lidocaine Patch
- Transdermal Hydrocolloid Placebo Patch (Placebo Comparator): Drug: Including placebo The intervention is the post-operative application of a hydrocolloid transdermal patch for women who have undergone Cesarean delivery.
  Interventions: Drug: Transdermal Hydrocolloid Placebo Patch

INTERVENTIONS:
Drug: Transdermal Lidocaine Patch — Transdermal Lidocaine Patch
  Other Names: Actavis US; NDC 0591-3525-30
  Arms: Transdermal Lidocaine Patch
Drug: Transdermal Hydrocolloid Placebo Patch — hydrocolloid placebo patches
  Other Names: DuoDerm; ConvaTec
  Arms: Transdermal Hydrocolloid Placebo Patch

SUMMARY:
This study will be a single-center, single blind, randomized controlled trial. The study will be conducted at UnityPoint-Health Meriter Hospital under investigators from the University of Wisconsin-Madison. Obstetric patients with prepregnancy obesity undergoing a Cesarean delivery at UnityPoint-Health Meriter will be eligible.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether transdermal lidocaine administered at the time of Cesarean delivery and for 12 hours postoperatively will reduce the total dose of opioids received. Our hypothesis is that a lidocaine patch will reduce the total dose of opioids received in the immediate 24 hours post-delivery. Secondary outcomes will include patient self-reported pain scores, patient-reported incidence of side effects, such as pruritis, development of objective complications, such as serious skin reactions (examples are acute generalized exanthematous pustolosis, Stevens-Johnson syndrome, and toxic epidermal necrolysis), hypersensitivity, nausea, and nervousness. Other outcomes collected will include length of stay, time to first rescue analgesic medication, total dose of opioids in 48 hours, use of supplemental oxygen during hospitalization, total dose of opioids during hospitalization, breastfeeding rates, both exclusive and in combination with formula use, amount of opioid prescribed at discharge and whether refills were requested or administered, rates of chronic pain at six weeks postpartum, and six week Edinburgh Depression Screen scores. Neonatal outcomes such as five-minute Apgar scores and development of adverse outcomes will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age greater than or equal to 18
* Prepregnancy body mass index greater than or equal to 30 kg/m2 or ≥35 kg/m2 at delivery if no prepregnancy/ early pregnancy weight available
* Singleton or multifetal pregnancy
* Able to receive neuraxial analgesia
* Planned/ scheduled Cesarean delivery OR non-urgent Cesarean delivery with adequate time to consider and consent to the study
* Gestational age greater or equal to 32 weeks

Exclusion Criteria:

* Known hypersensitivity to lidocaine or colloid patch (defined as a history of a reaction or allergy to lidocaine (injectable, intravenous, or transdermal) or hydrocolloid patch reported by patient or documented in the medical record) or patient report
* Contraindication to regional analgesia
* Positive urine drug screen at admission to the hospital, if ordered for clinical purposes.
* Current opioid use or opioid use disorder per patient report or documented in the medical record or the ePDMP (reviewed by PI 1-14 days prior to surgery)
* Chronic opioid use or opioid use disorder, either patient reported or documented in the medical record or the ePDMP (reviewed by PI 1-14 days prior to surgery), defined as opioid use on most days for >3 months
* Planned Cesarean hysterectomy (excluded due to anticipated blood loss and alternative pain control measures, possible prolonged intubation)
* Planned vertical midline incision
* Presence of renal dysfunction precluding the use of NSAIDs
* Ischemic heart disease, congestive heart failure, or cardiomyopathy of pregnancy
* Coagulopathy
* Planned discharge from the hospital less than 24 hours postpartum

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 66 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Antony, MD, Principal Investigator — UW-Madison Obstetrics and Gynecology
Locations (1):
- UnityPoint Health-Meriter Hospital, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Antony KM, Adams JH, Jacques L, Hetzel S, Chappell RJ, Gnadt SE, Tevaarwerk AJ. Lidocaine patches for postcesarean pain control in obese women: a pilot randomized controlled trial. Am J Obstet Gynecol MFM. 2021 Jan;3(1):100281. doi: 10.1016/j.ajogmf.2020.100281. Epub 2020 Nov 26. PMID 33451596

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 participants delivered prior to randomization, leaving 63 participants to start the trial
Period: Overall Study
Arm/Group | Transdermal Lidocaine Patch | Transdermal Hydrocolloid Placebo Patch
Started | 32 | 31
Participant Data Analyzed | 30 | 31
Completed | 30 | 31
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: baseline characteristics for participants who completed the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Transdermal Lidocaine Patch | Transdermal Hydrocolloid Placebo Patch | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 31 | 61
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (4.9) | 31.1 (5.2) | 31.83 (5.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 31 | 61
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 24 | 24 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 30 | 31 | 61
Ethnicity ( NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic | 3 | 3 | 6
  Non- Hispanic | 27 | 28 | 55

OUTCOME MEASURES:

1. Primary Outcome: Total Dose of Opioids Received in the First 24 Hours Following Cesarean
Description: The total dose of opioids received in the first 24 hours following Cesarean delivery measured as oral morphine equivalents. This total dose will be calculated for every subject in the study, and the average and standard deviation (or appropriate non-parametric values if the data is not normally distributed) will be compared between the subjects randomized to the intervention arm and the placebo arm of the study.
Time Frame: up to 24 hours
Measure: Mean (Standard Deviation); unit: MME, morphine milligram equivalents
Arm/Group | Transdermal Lidocaine Patch | Transdermal Hydrocolloid Placebo Patch
Number analyzed (Participants) | 30 | 31
MME, morphine milligram equivalents | 87 (35.8) | 83.9 (27.5)

2. Secondary Outcome: Post-operative Pain Score at 24 Hours Post-operatively
Description: The post-operative pain score at 24 hours post-operatively will be measured using the numeric rating scale (NRS), wherein subjects rate pain on a 0-10 scale (10 meaning the most pain and 0 meaning no pain). The median NRS score at 24 hours will be compared between the two groups.
Time Frame: up to 24 hours
Population: Median Pain Scores Overall and by Prepregancy and Delivery Body Mass Index (BMI)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Transdermal Lidocaine Patch | Transdermal Hydrocolloid Placebo Patch
Number analyzed (Participants) | 30 | 31
score on a scale
  Median Pain Score (0-10) | 3.0 [1.0 to 9.5] | 3.5 [1.0 to 7.0]
  Pre pregnancy BMI 30-39.9: number analyzed (Participants) | 20 | 20
  Pre pregnancy BMI 30-39.9 | 3.0 [2.0 to 3.2] | 3.0 [2.0 to 5.0]
  Prepregancy BMI >40: number analyzed (Participants) | 10 | 11
  Prepregancy BMI >40 | 4.0 [2.6 to 4.0] | 4.0 [3.0 to 5.0]
  Delivery BMI 30 -39.9: number analyzed (Participants) | 16 | 19
  Delivery BMI 30 -39.9 | 3.0 [2.4 to 4.0] | 3.0 [2.0 to 4.5]
  Delivery BMI >40: number analyzed (Participants) | 14 | 12
  Delivery BMI >40 | 3.0 [2.2 to 3.8] | 4.0 [3.0 to 5.2]

3. Other Pre Specified Outcome: Number of Participants With Opioid-related Side Effects
Description: Patient-reported opioid-related side effects include pruritis, constipation, nausea, and mental clouding.
  Definition: Patient reported side effects which will be reported as frequencies of occurrence. (These will be reported as dichotomous "Yes/No" outcomes for each side effect)
Time Frame: up to 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Transdermal Lidocaine Patch | Transdermal Hydrocolloid Placebo Patch
Number analyzed (Participants) | 30 | 31
Participants | 2 | 4

4. Other Pre Specified Outcome: Number of Participants With Complications of Lidocaine Use
Description: Complications of lidocaine use include local burning, nausea, dizziness, drowsiness, serious skin reactions such as blistering, confusion, blurred vision, ringing in the ears, and allergies and hypersensitivities.
  Definition: Patient reported side effects which will be reported as frequencies of occurrence. (These will be reported as dichotomous "Yes/No" outcomes for each side effect)
Time Frame: up to 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Transdermal Lidocaine Patch | Transdermal Hydrocolloid Placebo Patch
Number analyzed (Participants) | 30 | 31
Participants | 2 | 4

5. Other Pre Specified Outcome: Length of Hospital Stay
Description: Measured in hours from admission to time of discharge This will be measured in hours from the documented time of admission until discharge
Time Frame: up to 120 hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Transdermal Lidocaine Patch | Transdermal Hydrocolloid Placebo Patch
Number analyzed (Participants) | 30 | 31
hours | 75.5 [70.4 to 96.4] | 76 [71.3 to 91.7]

6. Other Pre Specified Outcome: Time to First Rescue Opioid Analgesic Medication
Description: Measured in minutes from arrival in the post-anesthesia care unit (PACU) until the first as needed opioid dose is administered. This will be recorded in minutes from the time of the surgery completion (surgery end time) until the first opioid analgesic medication is administered. Data in table is noted in hours.
Time Frame: up to 24 hours
Measure: Median (Full Range); unit: hours
Arm/Group | Transdermal Lidocaine Patch | Transdermal Hydrocolloid Placebo Patch
Number analyzed (Participants) | 30 | 31
hours | 1.4 [0.2 to 4.5] | 1.7 [0.2 to 4.0]

7. Other Pre Specified Outcome: Total Dose of Opioids Used in the First 48 Hours Post-operatively
Description: All opioid doses will be converted into oral morphine equivalents. This will be recorded as the total dose of opioids received in 48 hours following surgery calculated as oral morphine equivalents
Time Frame: up to 48 hours
Measure: Mean (Standard Deviation); unit: MME, morphine milligram equivalents
Arm/Group | Transdermal Lidocaine Patch | Transdermal Hydrocolloid Placebo Patch
Number analyzed (Participants) | 30 | 31
MME, morphine milligram equivalents | 149.3 (58.5) | 139.0 (48.9)

8. Other Pre Specified Outcome: Total Dose of Opioids During the Whole Hospitalization.
Description: All opioid doses will be converted into oral morphine equivalents. This will be recorded as the total dose of opioids received during the hospitalization (following surgery) calculated as oral morphine equivalents.
Time Frame: up to 120 hours
Measure: Median (Full Range); unit: MME, morphine milligram equivalents
Arm/Group | Transdermal Lidocaine Patch | Transdermal Hydrocolloid Placebo Patch
Number analyzed (Participants) | 30 | 31
MME, morphine milligram equivalents | 200 [0 to 448] | 192 [42 to 388]

9. Other Pre Specified Outcome: Number of Participants With Postoperative Complications
Description: Includes urinary tract infections, thromboembolic events, pneumonia, postpartum blood transfusions, falls, myocardial infarctions.
  These events will be reported as frequencies of occurrence. (These will be reported as dichotomous "Yes/No" outcomes for each side effect)
Time Frame: up to 120 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Transdermal Lidocaine Patch | Transdermal Hydrocolloid Placebo Patch
Number analyzed (Participants) | 30 | 31
Participants | 0 | 0

10. Other Pre Specified Outcome: Number of Opioid Pills Prescribed at Discharge
Description: The number of opioid pills prescribed at discharge
Time Frame: up to 72 hours
Measure: Mean (Standard Deviation); unit: Number of pills
Arm/Group | Transdermal Lidocaine Patch | Transdermal Hydrocolloid Placebo Patch
Number analyzed (Participants) | 30 | 31
Number of pills | 17.3 (9.0) | 16.0 (9.3)

11. Other Pre Specified Outcome: Neonatal Outcomes: Gestational Age at Delivery
Description: Gestational age at delivery will be recorded as weeks and days of gestation
Time Frame: up to 24 hours
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Transdermal Lidocaine Patch | Transdermal Hydrocolloid Placebo Patch
Number analyzed (Participants) | 30 | 31
weeks | 38.7 (1.7) | 38.85 (1.85)

12. Other Pre Specified Outcome: Dose Opioids (Measured in Total Morphine Milligram Equivalents (mg) of All Pills) Prescribed at Discharge
Description: Dose opioids (measured in total morphine milligram equivalents (mg) of all pills) prescribed at discharge
Time Frame: up to 72 hours
Measure: Mean (Standard Deviation); unit: MME (mg)
Arm/Group | Transdermal Lidocaine Patch | Transdermal Hydrocolloid Placebo Patch
Number analyzed (Participants) | 30 | 31
MME (mg) | 168.35 (120.4) | 154.10 (93.9)

ADVERSE EVENTS:
Time Frame: 6 weeks post partum
Arm/Group | Transdermal Lidocaine Patch | Transdermal Hydrocolloid Placebo Patch
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 2/30 | 0/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transdermal Lidocaine Patch (N=30) | Transdermal Hydrocolloid Placebo Patch (N=31)
Adverse Event ( not serious) (Surgical and medical procedures) | 1 (1) | 0 (0) — Seen in ER after initial hospital discharge for abdominal pain: resolved spontaneously. Outcome: Recovered without sequelae Severity: Mild SAE Category: "Other" AE Treatment: None Action taken: None Attribution: Relatedness: Unrelated
Adverse Event (not serious) (Surgical and medical procedures) | 1 (1) | 0 (0) — Delayed postpartum hemorrhage 6 weeks postpartum requiring D&C Outcome: Recovered without sequelae Severity: Moderate SAE Category: Other AE Treatment: Non-mediation treatment Action taken with study: None Attribution/ relatedness: Unrelated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-08): https://cdn.clinicaltrials.gov/large-docs/35/NCT03810235/Prot_SAP_001.pdf
  • Informed Consent Form (2019-02-13): https://cdn.clinicaltrials.gov/large-docs/35/NCT03810235/ICF_000.pdf